CLINICAL TRIAL: NCT02757495
Title: Can Caudal Dexmedetomidine Prevents Sevoflurane Induced Emergence Agitation in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ghada A.Kamhawy, lecturer of anesthesia,faculty of medicine, suez canal university, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: gkamhawy; Tarek F. Tammam (Other: Suez canal university)
Record Dates: First submitted 2016-04-13; First posted 2016-05-02 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Delayed Emergence From Anesthesia
Keywords: sevoflurane emergence agitation; caudal dexmedetomidine
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional (No Intervention): This will utilize the traditional method of performance of single dose caudal epidural block
- Caudal dexmedetomidine (Experimental): In this arm, single dose caudal epidural injection will be done patients in this arm will be given dexmedetomidine (precedex 100 µg/mL parenteral preparation (Hospira ® ) 2 µg/kg in 1 ml/kg bupivacaine 0.25%
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Single dose caudal epidural injection will be done using 25 G needle. patients of Group BD will be given dexmedetomidine (precedex 100 µg/mL parenteral preparation (Hospira ® ) 2 µg/kg in 1 ml/kg bupivacaine 0.25%,
  Other Names: Precedex
  Arms: Caudal dexmedetomidine

SUMMARY:
Emergence agitation (EA) is common phenomenon in pediatric patients undergoing general anesthesia by inhalation agents. The incidence of EA was reported to range from 18% to 80%. Sevoflurane now is the inhalational anesthetic agent of choice for pediatrics, Different strategies have been suggested to decrease the incidence and severity of EA. No gold standard technique for treating EA after sevoflurane anesthesia is currently available. The main question is can caudal dexmedetomidine be used for this purpose?

DETAILED DESCRIPTION:
The purpose of this prospective comparative randomized clinical study will be to compare the effects of caudal dexmedetomidine on EA in children undergoing lower abdominal operations under general sevoflurane anesthesia. In addition, characteristics of anesthesia recovery and incidence of adverse effects will be compare. A total of (48) children aged 1-5 years old, The American society of Anesthesiologists (ASA) physical status classification system between I-II of both sex who will be enrolled from April 2016 to April 2017 undergoing for lower abdominal surgeries will be included in the study. Patients will be randomized by computer-generated random numbers in a double blinded fashion to get enrolled into 2 equal groups: Group BD patients (n = 24) will be received single dose caudal epidural analgesia using dexmedetomidine with bupivacaine, whereas Group B patients (n = 24) will be received single dose caudal epidural analgesia with bupivacaine only. The dexmedetomidine used for this study will be prepared in a 1 ml syringe wrapped in aluminum foil by an investigator who will not be involved in the anesthesia process and another 1 ml syringe filled with saline will be prepared too.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-5 years old,
* The American society of Anesthesiologists (ASA) physical status classification system between I-II of both sex who will be enrolled from March 2015 to March 2016 undergoing for lower abdominal surgeries, e.g., hernia and perineal surgeries, e.g., undescended testis and hypospadius will be included in the study.

Exclusion Criteria:

* mental retardation, developmental delay, known allergy to any of the study drugs, congenital anomalies of spine, neurological or psychiatric illness that may be associated with improper communication, any signs of local infection in the sacrum region, any kind of cardiac conduction disorder, bleeding disorders, any previous cardiovascular disease and parental refusal.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Degree of Emergence Agitation will be evaluated-initial | upon awakening
  using the pediatric anesthesia emergence delirium scale (PAED), Patients will be considered agitated if they had a score of 16/20 or higher

SECONDARY OUTCOMES:
Incidence of emergence agitation at different time interval after surgery | 10 min ,20 min , 30 min and 60 min after surgery
  using the pediatric anesthesia emergence delirium scale (PAED), Patients will be considered agitated if they had a score of 16/20 or higher
Emergence time | immediately postoperative
  the time from the cessation of sevoflurane to the eye-opening will be noted.
Postoperative pain will be assessed, pain score will be observed and recorded at different time interval after surgery | immediately postoperative and every 4 hours in the first 24 hours
  Pain will be assessed by the pediatric observational 10-point scale "Face, Leg, Activity, Cry, Consolability (FLACC) pain score.
  Each category is scored on the 0-2 scale which results in a total score of 0-10.
  Assessment of Behavioural Score:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain Patients with pain score ≥4 will be given rescue analgesia

OTHER OUTCOMES:
Side-effect-bradycardia | intraoperatively and 24 hour postoperatively
  a heart rate less than 60 beats/min
Side-effect-hypotension | intraoperatively and 24 hour postoperatively
  Hypotension will be defined as a blood pressure below the 5th percentile for age and height
Side-effect-respiratory depression | intraoperatively and 24 hour postoperatively
  Respiratory depression will be defined as unable to maintain oxygen saturation of ≥ 95%.
Side-effect-urinary retention | intraoperatively and 24 hour postoperatively
  A urine output of less than 1 ml/kg/hr with a full bladder

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A. Kamhawy, Lecturer, Study Director — Suez Canal University
Locations (1):
- Suez canal University hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided